PRINCIPAL INVESTIGATOR: Steven Pavletic, MD

STUDY TITLE: A Phase I/II Trial of BMS-986253 in Myelodysplastic Syndromes

STUDY SITE: NIH Clinical Center

Cohort: Screening

Consent Version: 1/23/2023

# WHO DO YOU CONTACT ABOUT THIS STUDY?

**Principal Investigator:** Steven Pavletic, MD, MS

240-760-6174

pavletis@mail.nih.gov

#### KEY INFORMATION ABOUT THIS RESEARCH

This consent form describes a research study and is designed to help you decide if you would like to be a part of the research study.

You are being asked to take part in a research study at the National Institutes of Health (NIH). This section provides the information we believe is most helpful and important to you in making your decision about participating in this study. Additional information that may help you decide can be found in other sections of the document. Taking part in research at the NIH is your choice.

You are being asked to be screened for this study because you have been diagnosed with Myelodysplastic Syndromes (MDS).

This consent form requests your permission for us to determine your eligibility for our study involving treatment with BMS-986253 as a treatment for MDS.

The use of BMS-986253 in this study is considered investigational, which means that is has not been approved by the U.S. Food and Drug Administration (FDA) to treat MDS. However, the FDA has given us permission to use BMS-986253 in this study.

There are other drugs that may be used to treat your disease, and these can be prescribed/given by your regular doctor, even if you are not in this study. Some examples include: other DNMTi therapy such as azacitidine or decitabine, other oral treatments such as lenalidomide, or drugs that would not treat the disease directly but may help improve your blood counts and overall symptoms, such as erythropoietin stimulating agents.

The goal of this study is to determine if BMS-986253 is a safe and effective treatment for Myelodysplastic Syndromes (MDS). The first phase of this research study will determine the largest dose of BMS-986253 that can be safely given to patients with MDS. The second phase of this research study will determine how well patients with MDS respond to BMS-986253.

This consent is for "screening." We would like to "screen" you to find out if you are able to take part in this study, and this could mean that we will use samples from procedures you have undergone at home or in the Clinical Center.

## PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (2)

Version Date: 1/23/2023




If you decide to be screened for this study, here are some of the most important things that you should know that will happen.

We will first do some basic tests to make sure you qualify for the trial. These basic tests involve blood tests, images, and physical exams, etc. Other tests are described further on in this consent form. It is important that you read these.

There is a chance that you may experience side effects from the tests to be done (for example: pain from blood draws where the needle enters the skin).

You will not benefit from this screening evaluation.

You may choose not to be tested for eligibility or to have any other studies done.

You are free to stop participating in the trial at any time.

The remaining document will now describe the research study in more detail. This information should be considered before you make your choice. Members of the study team will talk with you about the information in this document. Some people have personal, religious, or ethical beliefs that may limit the kinds of medical or research interventions in which they would want to participate. Take the time you need to ask any questions and discuss this study with NIH staff, and with your family, friends, and personal health care providers.

# IT IS YOUR CHOICE TO TAKE PART IN THE STUDY

You may choose not to take part in this study for any reason. If you join this study, you may change your mind and stop participating in the study at any time and for any reason. In either case, you will not lose any benefits to which you are otherwise entitled. However, to be seen at the NIH, you must be taking part in a study or are being considered for a study. If you do choose to leave the study, please inform your study team to ensure a safe withdrawal from the research.

#### WHY IS THIS STUDY BEING DONE?

The purpose of the phase I portion of this study is to test the safety of BMS-986253 at different doses to find out what effects, if any, it has on participants with MDS to determine the recommended dose for the phase 2 part of the trial. The purpose of the phase II portion of the study is to determine the response rate to BMS-986253.

You are being asked to join this study because you have been diagnosed with MDS.

You may not be eligible for our study with BMS-986253 for several reasons, such as the presence of certain other diseases, infections, or blood counts which are not in the correct range.

In order to see if you are eligible to take part in the research, we are asking you to first take part in this screening portion of the study.

## WHAT WILL HAPPEN DURING THE STUDY?

During the screening period, your doctor will make sure you are able to take part in the study.

You will be asked questions about your medical history, and prescription or non-prescription medications you take or have taken, the history or your disease and how well you are able to care for yourself.

## PATIENT IDENTIFICATION

**Consent to Participate in a Clinical Research Study** 

NIH-2977 (4-17)

File in Section 4: Protocol Consent (2)




You will undergo the following tests/assessments to see whether you are able to take part in the study:

- Medical history
- Physical examination
- Laboratory evaluations
- ECG

# Required screening assessments:

During your screening period you will:

- Visit the NIH Clinical Center to answer questions about your medical history
- Answer questions about how well you are able to take care of yourself
- List any prescriptions or non-prescription medicines you have taken
- Discuss the history of you MDS and any other medicines you have taken for the MDS.
- Have a physical exam (including height and weight)
- Have your temperature, blood pressure, breathing rate, oxygen saturation, and heart rate monitored
- Have an electrocardiogram (ECG) a test to show how well your heart is working
- Have blood samples taken to check your blood counts, blood minerals, liver and kidney function, and to screen for certain viruses (approximately 3 tablespoons).
- A bone marrow biopsy may be performed to confirm your diagnosis of MDS if unable to confirm by obtaining an outside bone marrow sample
- If you are a female who can have children, a urine and/or blood pregnancy test will be done. If urine test if positive, it will be confirmed with a blood test (approximately 1 teaspoon). The results of the blood test must be negative for you be allowed to participate in the study.

As part of this study, we will test you for infection with HIV, the virus that causes AIDS. If you are infected with HIV, you will not be able to take part in this study. We will tell you what the results mean, how to find care, how to avoid infecting others, how we report HIV infections, and the importance of informing your partners at possible risk because of your HIV infection.

If the tests or if your answers show that you are not able to take part in the study, you will not be allowed to continue. Your study doctor will discuss other care options with you.

If you are able to take part in the study, your study doctor will assign you to a specific group.

You will also be assigned to a specific subgroup to receive either BMS-986253 monotherapy or in combination with a DNMTi (decitabine and cedazuridine). Your study doctor will inform you of your treatment plan.

# HOW LONG WILL THE STUDY TAKE?

If you agree to take part in this screening, your involvement will last for the length of time to see if you are eligible to take part in the research treatment phase of the study. The length of time may range anywhere from a couple weeks to several months. You will be required to come to NIH at least one-time during screening and the visit may last anywhere from 1 to 14 days.

## PATIENT IDENTIFICATION

**Consent to Participate in a Clinical Research Study** 

NIH-2977 (4-17)

File in Section 4: Protocol Consent (2)




## HOW MANY PEOPLE WILL PARTICIPATE IN THIS STUDY?

As not all persons screened will be eligible for study therapy, up to 200 patients will be enrolled in order to treat about 93 subjects on the study.

## WHAT ARE THE RISKS AND DISCOMFORTS OF BEING IN THE STUDY?

Listed below are possible risks and discomforts with being in this screening part of the study:

# **Blood samples**

Side effects of repeated blood sampling depend in part on how the blood is drawn. If through an intravenous catheter, risks include contamination of the catheter which could result in a serious blood stream infection, requiring admission to the hospital and giving you antibiotics through the vein; if blood is drawn through a needle into your skin, side effects could include pain and bruising in the area where the blood was drawn. Other side effects can include bruising, redness, discomfort or bleeding at the site of the needle stick, and possible lightheadedness, or rarely, fainting. If you have too much blood taken over a prolonged period, your red blood cell count may drop (this is called "anemia"). As a precaution, we will check your red blood cell level, and give you an iron treatment or a blood transfusion if needed. Approximately 3.5 tablespoons of blood may be drawn for this screening process.

# Electrocardiogram

Other than possibly experiencing some minor skin irritation from the electrodes, there are no anticipated risks related to completing the electrocardiogram and/or the echocardiogram.

# **Bone Marrow Aspiration/Biopsy**

The bone marrow aspiration and biopsy may cause pain, bruising, bleeding, and infection. Soreness near the site may last for a couple of days after the procedure. You may have more pain, risk of bleeding and bruising if you complete both aspiration and biopsy rather than just the aspiration. If your pain is severe or you develop a fever, please contact the study team immediately.

# What are the risks related to pregnancy?

If you are able to become pregnant, we will ask you to have a pregnancy test before starting this study. You must use effective birth control methods prior to study entry and try not to become pregnant while participating in this study <u>or</u> during study treatment, and for 6 months after you finish study treatment. If you become pregnant, there may be unknown risks to the fetus or unborn child, or risks that we did not anticipate. There may be long-term effects of the treatment being studied that could increase the risk of harm to a fetus. You must tell the study doctor if your birth control method fails while you are in the study. If you think or know you have become pregnant while participating in this research study, please contact the study team as soon as possible. If you plan to become pregnant in the future, please discuss with the study team how long you need to wait before becoming pregnant after completing the study.

If you are a sexually active person with a partner able to become pregnant, it is important that your partner not become pregnant during your participation in this study <u>or</u> during study treatment, and for 6 months after you finish study treatment. There may be unknown risks to a fetus or risks we

## PATIENT IDENTIFICATION

**Consent to Participate in a Clinical Research Study** 

NIH-2977 (4-17)

File in Section 4: Protocol Consent (2)




did not anticipate. You and your partner must agree to use birth control if you want to take part in this study. If you think your partner has become pregnant during your participation in this study, please contact the study team as soon as possible. If you and your partner plan for your partner to become pregnant after your participation in this study, please discuss this with the study team.

# **Privacy Risks Associated with Genetic Testing**

It may be possible that genetic information from you could be used by law enforcement agencies or other entities to identify you or your blood relatives

# PSYCHOLOGICAL OR SOCIAL RISKS ASSOCIATED WITH RETURN OF INCIDENTAL OR SECONDARY FINDINGS

As part of the research study, it is possible that you could learn that you have genetic risks for another disease or disability. This may be upsetting and, depending on what you learn, might create a need to make challenging decisions about how to respond.

Although your genomic information is unique to you, you share some genomic similarities with your children, parents, brothers, sisters, and other blood relatives. Therefore, learning your research results could mean something about your family members and might cause you or your family distress. Before joining the study, it may be beneficial to talk with your family members about whether and how they want you to share your results with them.

#### PROTECTIONS AGAINST MISUSE OF GENETIC INFORMATION

This study involves genetic testing on samples. Some genetic information can help predict future health problems of you and your family and this information might be of interest to your employers or insurers. The Genetic Information Nondiscrimination Act (GINA) is a federal law that prohibits plans and health insurers from requesting genetic information or using genetic information. It also prohibits employment discrimination based on your health information. However, GINA does not address discrimination by companies that sell life insurance, disability insurance, or long-term care insurance. GINA also does not protect you against discrimination based on an already-diagnosed condition or disease that has a genetic component.

## WHAT ARE THE BENEFITS OF BEING IN THE STUDY?

You will not benefit from this screening evaluation; however, this will determine if you are eligible to participate in the clinical trial.

# Are there any potential benefits to others that might result from the study?

In the future, other people might benefit from this study because the knowledge gained from this study may be used to help treat others who have MDS.

## WHAT OTHER OPTIONS ARE THERE FOR YOU?

You may choose not to be tested for eligibility or to have any other studies done.

## DISCUSSION OF FINDINGS

## New information about the study

If we find out any new information that may affect your choice to participate in this study, we will get in touch with you to explain what we have learned. This may be information we have

## PATIENT IDENTIFICATION

**Consent to Participate in a Clinical Research Study** 

NIH-2977 (4-17)

File in Section 4: Protocol Consent (2)




learned while doing this study here at the NIH or information we have learned from other scientists doing similar research in other places.

## Return of research results

The results from the evaluations for this screening will be reported to you. You will be informed at that time if you are eligible for the main study.

## EARLY WITHDRAWAL FROM THE STUDY

Your doctor may decide to stop your screening evaluation for the following reasons:

- if he/she believes that it is in your best interest
- if you are ineligible for the study
- if you become pregnant
- if new information shows that another treatment would be better for you
- if the study is stopped for any reason

If your evaluation is stopped, you will be informed of the reason screening is being stopped. You can stop taking part in the study at any time. However, if you decide to stop taking part in the study, we would like you to talk to the study doctor and your regular doctor first.

If you decide at any time to withdraw your consent to participate in the trial, we will not collect any additional medical information about you. However, according to FDA guidelines, information collected on you up to that point may still be provided to our collaborators or designated representatives.

# STORAGE, SHARING AND FUTURE RESEARCH USING YOUR SPECIMENS AND DATA

# Will your specimens or data be saved by the study team for use in other studies?

As part of this study, we are obtaining specimens and data from you. We plan to store and use these specimens and data for studies other than the one described in this consent form that are going on right now, as well as studies that may be conducted in the future. The specimens and data will be kept in a way that we will still know that they came from you (i.e., they will be identifiable to us). If we use your identifiable specimens or data for future research, our study will be reviewed and approved by an Institutional Review Board who will make sure that we are protecting your confidentiality. These future studies might help us better understand myelodysplastic syndromes, or other diseases or conditions. This could include studies to develop other research tests, treatments, drugs, or devices, that may lead to the development of a commercial product by the NIH and/or its research or commercial partners. There are no plans to provide financial compensation to you if this happens. Also, it is unlikely that we will learn anything from these studies that may directly benefit you.

I give permission for my identifiable specimens and data to be stored and used by the study team for future studies as described above.

| Yes | No |
|---------|---------|
| Initial | Initial |

PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (2) Version Date: 1/23/2023




# Will your specimens or data be shared with other researchers for use in other studies?

We may share your specimens and data with other researchers. The other researchers may be doing studies in similar areas to this study or in other unrelated areas. These researchers may be at NIH, other research centers and institutions, or commercial entities.

If we do share your specimens or data, we will know that the specimens and data came from you. However, the other researchers will not know that they came from you (i.e., they will be deidentified).

I give permission for my de-identified specimens and data to be shared with and used by other researchers for future studies.

| Yes | | No |
|---------|---------|----|
| Initial | Initial | |

In some cases, it may help other researchers to know that the specimens or data were collected from you (i.e., they will have your identifiers). If we share your identity with other researchers, their study will be reviewed and approved by an Institutional Review Board who will make sure that the study team is protecting your confidentiality.

I give permission for my identifiable specimens and data to be shared with and used by other researchers for future studies.

| Y | es | | No |
|---------|----|---------|----|
| Initial | | Initial | |

In addition to the planned use and sharing described above, we might remove any labels from your specimens and data that might identify you (i.e., anonymize them), and use them or share them with other researchers for future studies at the NIH or other places. When we or the other researchers use your anonymized specimens and data for these projects, there will be no way to know that they came from you. We want to make sure that you understand that this is a possibility if you participate in this study. Once we do this, we would not be able to remove your specimens or data from these studies or prevent their use in future research studies because we would not be able to tell which specimens or data belong to you.

## Can you change your mind about use and sharing for future research?

If you change your mind and do not want us to store and use your specimens and data for future studies, you should contact the study team. We will do our best to comply with your request but cannot guarantee that we will always be able to destroy your specimens and data. For example, if some research with your specimens and data is already complete, the information from that research may still be used. Also, if the specimens and data have been shared already, it might not be possible to withdraw them.

## PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (2)




# Will your genomic data be shared outside of this study?

As part of this research study, we will put your genomic information in a large database for broad sharing with the research community. These databases are commonly called data repositories. The information in this database will include, but is not limited to, genetic information, race, ethnicity and sex. If your information is placed in one of these repositories, it will be labeled with a code (not with your name or other information that could be used to easily identify you), and only qualified researchers will be able to access it. These researchers must receive permission from individuals or committees with the authority to determine whether these researchers can access the data. Before receiving the data, the researchers must promise that they will not attempt to re-identify the subjects whose data they will receive.

Genomic summary information about all of the participants included in this study (including you) is being placed in a database and will be available through open access. This information will help the researchers understand if some genetic patterns are more common than others among the subjects who participated in the study. The researchers and non-researchers will be able to access genomic summary information about all the participants included in the study, or summary information combined from multiple studies, without applying for permission. The risk of anyone identifying you based on this information is very low.

# How long will your specimens and data be stored by the NIH?

Your specimens and data may be stored by the NIH indefinitely.

# Risks of storage and sharing of specimens and data

When we store your specimens and data, we take precautions to protect your information from others that should not have access to it. When we share your specimens and data, we will do everything we can to protect your identity, for example, when appropriate, we remove information that can identify you. Even with the safeguards we put in place, we cannot guarantee that your identity will never become known or that no one will gain unauthorized access to your information. New methods may be created in the future that could make it possible to re-identify your specimens and data.

#### **PAYMENT**

# Will you receive any type of payment for taking part in this study?

You will not receive any payment for taking part in this study.

## REIMBURSEMENT

# Will you receive reimbursement or direct payment by NIH as part of your participation?

On this study, the NCI will reimburse the cost for some of your expenses such as those for hotel, travel, meals. Some of these costs may be paid directly by the NIH and some may be reimbursed after you have paid. The amount and form of these payments are determined by the NCI Travel and Lodging Reimbursement Policy. You will be given a summary of the policy which provides more information.

## PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (2)




If your travel to the NIH Clinical Center (e.g. flight, hotel) is arranged and paid for by the NIH, the agency making the reservations and their representatives will have access to your identifiable information.

# **COSTS**

# Will taking part in this research study cost you anything?

NIH does not bill health insurance companies or participants for any research or related clinical care that you receive at the NIH Clinical Center.

• If some tests and procedures are performed outside the NIH Clinical Center, you may have to pay for these costs.

# **CONFLICT OF INTEREST (COI)**

The NIH reviews NIH staff researchers at least yearly for conflicts of interest. This process is detailed in a COI Guide. You may ask your research team for a copy of the COI Guide or for more information. Members of the research team who do not work for NIH are expected to follow these guidelines or the guidelines of their home institution, but they do not need to report their personal finances to the NIH.

The NIH and the research team for this study are using BMS-986253 developed by Bristol Myers Squibb through a collaboration between your study team and the company. The company also provides financial support for this study.

# CLINICAL TRIAL REGISTRATION AND RESULTS REPORTING

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

# CONFIDENTIALITY PROTECTIONS PROVIDED IN THIS STUDY

## Will your medical information be kept private?

We will do our best to make sure that the personal information in your medical record will be kept private. However, we cannot guarantee total privacy. Organizations that may look at and/or copy your medical records for research, quality assurance, and data analysis include:

- The NIH and other government agencies, like the Food and Drug Administration (FDA), which are involved in keeping research safe for people.
- National Institutes of Health Intramural Institutional Review Board
- The study Sponsor (Center for Cancer Research) or their agent(s)
- Qualified representatives from Bristol Myers Squibb, the pharmaceutical company who produces BMS-986253.

The researchers conducting this study and the NIH follow applicable laws and policies to keep your identifying information private to the extent possible. However, there is always a chance that, despite our best efforts, your identity and/or information about your participation in this research may be inadvertently released or improperly accessed by unauthorized persons.

## PATIENT IDENTIFICATION

**Consent to Participate in a Clinical Research Study** 

NIH-2977 (4-17)

File in Section 4: Protocol Consent (2)




In most cases, the NIH will not release any identifiable information collected about you without your written permission. However, your information may be shared as described in the section of this document on sharing of specimens and data, and as further outlined in the following sections.

Further, the information collected for this study is protected by NIH under a Certificate of Confidentiality and the Privacy Act.

# **Certificate of Confidentiality**

To help us protect your privacy, the NIH Intramural Program has received a Certificate of Confidentiality (Certificate). With this certificate, researchers may not release or use data or information about you except in certain circumstances.

NIH researchers must not share information that may identify you in any federal, state, or local civil, criminal, administrative, legislative, or other proceedings, for example, if requested by a court.

The Certificate does not protect your information when it:

- 1. is disclosed to people connected with the research, for example, information may be used for auditing or program evaluation internally by the NIH; or
- 2. is required to be disclosed by Federal, State, or local laws, for example, when information must be disclosed to meet the legal requirements of the federal Food and Drug Administration (FDA);
- 3. is for other research;
- 4. is disclosed with your consent.

The Certificate does not prevent you from voluntarily releasing information about yourself or your involvement in this research.

The Certificate will not be used to prevent disclosure to state or local authorities of harm to self or others including, for example, child abuse and neglect, and by signing below you consent to those disclosures. Other permissions for release may be made by signing NIH forms, such as the Notice and Acknowledgement of Information Practices consent.

# **Privacy Act**

The Federal Privacy Act generally protects the confidentiality of your NIH medical information that we collect under the authority of the Public Health Service Act. In some cases, the Privacy Act protections differ from the Certificate of Confidentiality. For example, sometimes the Privacy Act allows release of information from your record without your permission, for example, if it is requested by Congress. Information may also be released for certain research purposes with due consideration and protection, to those engaged by the agency for research purposes, to certain federal and state agencies, for HIV partner notification, for infectious disease or abuse or neglect reporting, to tumor registries, for quality assessment and medical audits, or when the NIH is involved in a lawsuit. However, NIH will only release information from your medical record if it is permitted by both the Certificate of Confidentiality and the Privacy Act.

## POLICY REGARDING RESEARCH-RELATED INJURIES

The NIH Clinical Center will provide short-term medical care for any injury resulting from your participation in research here. In general, no long-term medical care or financial compensation for

PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17) File in Section 4: Protocol Consent (2)

Version Date: 1/23/2023 Page **10** of **12** 



research-related injuries will be provided by the NIH, the NIH Clinical Center, or the Federal Government. However, you have the right to pursue legal remedy if you believe that your injury justifies such action.

# PROBLEMS OR QUESTIONS

If you have any problems or questions about this study, about your rights as a research participant, or about any research-related injury, contact the Principal Investigator, Steven Pavletic, MD, pavletis@mail.nih.gov, 240-760-6174. Other researchers you may call are: Noa Holtzman, MD, at 240-858-3224. You may also call the NIH Clinical Center Patient Representative at 301-496-2626, or the NIH Office of IRB Operations at 301-402-3713, if you have a research-related complaint or concern.

## **CONSENT DOCUMENT**

Please keep a copy of this document in case you want to read it again.

PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (2)




| Adult Research Participant: I have read the explanation about this study and have been given the opportunity to discuss it and to ask questions. I consent to participate in this study. | | |
|---|---|---|
| Signature of Research Participant | Print Name of Research Participant | Date |
| Investigator: | | |
| Signature of Investigator | Print Name of Investigator | Date |
| Witness should sign below if either: 1. A short form consent process has been used to enroll a non-English speaking subject or 2. An oral presentation of the full consent has been used to enroll a blind or illiterate subject | | |
| Signature of Witness | Print Name of Witness | Date |
| NIH ADMINISTRATIVE SECTION TO BE COMPLETED REGARDING THE USE OF AN INTERPRETER: An interpreter, or other individual, who speaks English and the participant's preferred language facilitated the administration of informed consent and served as a witness. The investigator obtaining consent may not also serve as the witness. An interpreter, or other individual, who speaks English and the participant's preferred language facilitated the administration of informed consent but did not serve as a witness. The name or ID code of the person providing interpretive support is: | | |

PATIENT IDENTIFICATION

**Consent to Participate in a Clinical Research Study** 

NIH-2977 (4-17)

File in Section 4: Protocol Consent (2)


